CLINICAL TRIAL: NCT02803515
Title: HSP90 as a Predictive Marker of the Response to Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in the Treatment of Peritoneal Carcinomatosis From Ovarian Origin.
Brief Title: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) : Predictive Marker and Mechanism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOI-11
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Peritoneal Carcinomatosis
Keywords: intra peritonal chemo hyperthermia; peritoneal carcinomatosis; ovarian cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with HIPEC (Experimental)
  Interventions: Biological: peripheral venous blood samples
- Patient without HIPEC (Sham Comparator)
  Interventions: Biological: peripheral venous blood samples

INTERVENTIONS:
Biological: peripheral venous blood samples — peripheral venous blood samples measured preoperatively and postoperatively HIPEC (Day 1, day 3 and day 5 postoperative)

SUMMARY:
Peritoneal carcinomatosis (PC) is the stage III of the FIGO ovarian cancer staging. It corresponds to an advanced stage with a relative 5 year survival rate of 52%. The multimodal treatment approach combines neoadjuvant chemotherapy, cytoreductive surgery of macroscopic lesions, and hyperthermic intraperitoneal chemotherapy (HIPEC). It has significantly improved survival rate in patients with ovarian PC and decreased recurrence and mortality rate by 21%. The efficacy of HIPEC is based on chemotherapy potentiated by the hyperthermia (43°). However, the cellular mechanisms involved are not fully understood, but they include cell death pathways and heat shock proteins (Hsp70 and Hsp90). RICCI et al. showed, based on pre-clinical models, that the efficacy of HIPEC was partly due to the overexpression and exposure of HSP90 on the cell surface leaded to an anti-cancer immune response. The aims of this study are to validate these findings in tissue samples of patients with ovarian PC. We will constitute a bank of isolated tumor samples before and after HIPEC and measure postoperative HSP90 serum levels in order to establish if they are predictive of a response. HSPs expression on the cancer cell surface will be determined by flow cytometry. Forty-four patients will be included. Elucidating the underlying mechanisms of HIPEC will broaden therapeutic possibilities including the use of new immunotherapy. The multimodal approach could improve the efficacy of HIPEC with a minimal systemic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Females over 18 years.
* Indication of Hyperthermic Intra Peritoneal Chemotherapy (HIPEC) for peritoneal carcinomatosis from ovarian origin
* Obtaining written informed consent and signed for participation in the study and conservation of samples taken.
* Affiliation to a social security scheme.

Non-inclusion criteria

* Major patients protected by law or deprived of liberty.
* Patients pregnant women in labor or breastfeeding.
* Refusal of participation
* Another cause of peritoneal carcinomatosis

Exclusion Criteria:

* consent withdrawn

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
Changes in serum levels of HSP90 and 70 on peripheral venous samples. | basal levels (preoperatively), postoperatively HIPEC (Day 1, day 3 and day 5 postoperative)
  Changes in serum levels of HSP90 and 70 postoperatively HIPEC (Day 1, day 3 and day 5 postoperative) compared to basal levels measured preoperatively on peripheral venous samples. Patients who had HIPEC will be compared with patients overturned on early intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc BEREDER, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Digestive department - Archet hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided